CLINICAL TRIAL: NCT03109717
Title: Structural and Functional Connectivity of Brainstem Monoamine Pathways in Treatment Resistant Depression
Acronym: MAOI
Status: Completed | Type: Observational
Sponsor: Kathryn O'Connor (Other)
Responsible Party: Sponsor-Investigator, Kathryn O'Connor, Administrator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 15-1372
Record Dates: First submitted 2017-03-01; First posted 2017-04-12 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Treatment Resistant Depression
Keywords: Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Monoamine Oxidase Inhibitors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Resistant Depression: Screened for eligibility using several psychiatric assessments. If qualifies to participate in the study, will have to stop any antidepressants that they are taking to prepare for the use of Monoamine Oxidase Inhibitor(MAOI). After a two week washout period, subjects will have an fMRI and will be started on a MAOI. Then be followed for 8 weeks, part of routine care.
  Interventions: Drug: Monoamine Oxidase Inhibitor (MAOI)
- Healthy Control: Screen for eligibility, then MRI.

INTERVENTIONS:
Drug: Monoamine Oxidase Inhibitor (MAOI) — Monoamine Oxidase Inhibitor
  Other Names: Monoamine Oxidase Inhibitor
  Groups: Treatment Resistant Depression

SUMMARY:
Study TRD subjects' resistance to at least 2 different antidepressants, we hypothesize that because of their significant depression and treatment resistant status they are most likely to exhibit BSMN pathway abnormalities.

DETAILED DESCRIPTION:
Potential subjects will be identified during clinical visits. If a patient qualifies to participate in the study they will have to stop any antidepressants that they are taking to prepare for the use of MAOIs. After a two week washout period, subjects will have an fMRI and will be started on a MAOI. They will then be followed up for 8 weeks, which is routine and considered standard care.

ELIGIBILITY:
Inclusion Criteria - TRD:

1. age: 18 - 65 yrs.;
2. satisfy criteria for DSM-IV major depressive disorder (MDD);
3. 17-item Hamilton Depression Rating Scale (17-item HDRS) score > 18;
4. treatment resistance depression as defined as report of inadequate response (patient report of minimal improvement or nonresponse) despite past treatment with at least 2 different classes of antidepressants acting on the 5-HT and/or DA monoamine systems(except MAOIs) (as determined with the Antidepressant Treatment History Form (ATHF)20 with score of >3 on each of the items and verified by medical records if available);
5. able to give informed consent;
6. no use of alcohol in the past 1 week and negative urine toxicology screen;
7. MAOI treatment indicated as assessed by an independent psychiatrist not affiliated with the study;
8. voluntary consent to treatment with an MAOI after reviewing all other options and agree to follow safeguards and precautions during treatment.

Inclusion criteria for healthy subjects

1. ages 18-65 years and ability to give voluntary informed consent;
2. no history of psychiatric illness or substance abuse or dependence;
3. no significant family history of psychiatric or neurological illness;
4. not currently taking any prescription or centrally acting medications; no use of alcohol in the past 1 week;
5. and no serious medical or neurological illness.

Exclusion Criteria - TRD:

1. schizophrenia, schizoaffective or primary anxiety disorder;
2. serious medical or neurological illness;
3. history of significant head injury;
4. on fluoxetine treatment;
5. on lithium or have received ECT or rTMS in the last 3 months to avoid long-term effects of such medications;
6. substance or alcohol dependence in the past 6 months or substance abuse in the past 3 months;
7. unable to give informed consent.

Exclusion criteria for both groups:

1. pregnant or breast-feeding;
2. metallic implants or other contraindication to MRI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Treatment Resistant Depression and Healthy Controls
Sampling Method: Non-Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-11 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
Brainstem Structural Connectivity (Sc) | 2 years
  Localize BSMN and measure pathway Sc using diffusion imaging to differentiate between TRD and HC. BSMN can be localized using diffusion imaging, and pathways projecting from BSMN to known targets can be identified. Methods have been developed to localize these nuclei via a combination of diffusion imaging and anatomic imaging. We will identify these nuclei and track their projections to known targets, giving rise to the VTA-NAcc, VTA-AMYG, RN-AM and RN-sgACC pathways. Probabilistic fiber tracking between these nodes will be used to determine a measure of pathway strength.
Brainstem Functional Connectivity (Fc) | 2 years
  Measure BSMN pathway Fc to differentiate between TRD and HC. BSMN associated with different neuromodulators, e.g. the VTA and RN, will be associated with distinct functional networks which will be abnormal in TRD compared to HCs.

OTHER OUTCOMES:
17-item Hamilton Depression Rating Scale | 2 years
  Compare baseline and end of study Hamilton depression Rating scale and imaging correlations.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Anand, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No